CLINICAL TRIAL: NCT05114382
Title: An Evaluation of the Safety and Performance of the CathVision Cube® System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CathVision ApS (Industry)
Collaborators: TRIQ GROUP Wherry & Klaffke GbR (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-00003
Record Dates: First submitted 2021-08-16; First posted 2021-11-10 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-11

CONDITIONS: Cardiac Arrhythmia
Keywords: atrial fibrillation; pulmonary vein isolation; radiofrequency; cryo balloon; ablation; software
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A prospective, single center, open-label, single arm study to evaluate the safety and technical performance of the CathVision Cube® system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A prospective, multi-center, open-label, single arm study (Other): Patients undergoing assessment and ablation of cardiac arrhythmiast. who are scheduled for an electrophysiology (EP) procedure and meet all inclusion criteria will be enrolled in the study and undergo the EP procedure. Intracardiac signals will be passively recorded using the CathVision Cube® System in parallel with the commercial (CE marked) EP recording system for post procedure evaluation. The investigational device will not be used for direct clinical care decisions or therapy. The EP procedure will be guided by the study site Standards Of Care.
  Interventions: Procedure: EP Procedure

INTERVENTIONS:
Procedure: EP Procedure — Intracardiac signals will be passively recorded using CathVision Cube® System in parallel with the commercial (CE marked) EP recording system during a scheduled electrophysiology procedure
  Other Names: electrophysiology procedure

SUMMARY:
The primary objective is to evaluate the safety and technical performance of the CathVision Cube® System. The secondary objective is to benchmark the intracardiac electrogram signal quality compared to commercially available systems in patients undergoing assessment and ablation of cardiac arrhythmias.

DETAILED DESCRIPTION:
A prospective, single center, open-label, single arm study to evaluate the safety and technical performance of the CathVision Cube® system.

Patients undergoing assessment and ablation of cardiac arrhythmias, by Electro Physiology (EP) procedure, and who meet all inclusion criteria will be enrolled in the study and undergo the EP procedure. Intracardiac signals will be passively recorded using the CathVision Cube® System in parallel with a commercial (CE marked) EP recording system and later compared and evaluated. The investigational device will not be used for direct clinical care decisions or therapy. The EP procedure will be guided by the study site Standards Of Care.

ELIGIBILITY:
Inclusion Criteria:

* Patient indicated by investigator for catheter ablation or diagnostic electrophysiology procedure.
* Male or non-pregnant female aged ≥18 years. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days prior to index procedure.
* Able and willing to directly provide informed consent.

Exclusion Criteria:

* Patient inability to understand or refusal to sign informed consent.
* Pregnant or nursing patients and those who plan pregnancy in the period up to 1 month following the index procedure.
* Current participation in another investigational drug or device study that interferes with this study.
* Patient is a prisoner.
* Patients who in the opinion of the physician are not candidates for this study. Prior atrial septal defect (ASD) or patent foramen ovale (PFO) closure with a device using a transcatheter percutaneous approach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Freedom from major adverse events, evaluated at hospital discharge. | From EP procedure to hospital discharge is 1 day
  Freedom from major adverse events, evaluated at hospital discharge
Recording low-voltage electrograms | Duration of the EP procedure can take up to 6 hours
  Recording low-voltage electrograms under 20uV amplitude
The Primary Performance endpoint of study will be evaluated as technical success of CathVision Cube® system to collect and record intracardiac signals during EP procedures | Duration of the EP procedure can take up to 6 hours
  Logging time for arrhythmia termination / block
Compatibility of Cube System with commercially available 3D mapping system | Duration of the EP procedure can take up to 6 hours
  Assessing compatibility of Cube System with commercially available 3D mapping system with available intracardiac catheters. Compatibility is assessed by that the Cube System does not introduce a visual detectable distortion on the commercial available 3D mapping systems

CONTACTS AND LOCATIONS:
Overall Officials: Josef Kautzner, Prof., Principal Investigator — IKEM, Prague, Czech Republic; Peter K Jacobsen, MD, DMSc, Principal Investigator — Righospitalet, Copenhagen, Denmark
Locations (2):
- IKEM, Institue of Clinical and Experimental Medicine, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No